CLINICAL TRIAL: NCT03915587
Title: Bedside Resources to Gauge Intravascular Volume Status in Hypovolemic Infants in the Operating Room
Brief Title: Bedside Resources to Gauge Intravascular Volume Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-2513
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hypovolemia; Craniosynostoses
MeSH Terms: conditions — Hypovolemia; Craniosynostoses

STUDY DESIGN:
Intervention Model Description: Single arm prospective trial which will define two groups
Masking Description: As these devices are experimental in this patient population, anesthesiologists will be blinded to hemodynamic data generated by the CardioQ-EDM, bedside ultrasound, and CipherOx CRI. If data is needed in an emergent setting, the subject will be excluded from analysis. Although recorded measurements from the Cardio-Q EDM monitor will be visible to the study team, IVC measurements will be stored and calculated post-hoc by a co-investigator blinded to whether or not the subject is or is not fluid responsive. Additionally, a trained statistician not involved in data collection will be paid for analysis. It should also be noted at Dr. Steven Moulton is a paid officer of CipherOx but will not be involved in the data collection and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fluid Challenge (Other): After defining fluid responders from non-responders in this single arm prospective trial, we will compare the predictive utility of non-invasive devices such as the CipherOx-CRI and IVC CI to currently employed indices (heart rate, systolic blood pressure, urine output and pulse pressure variability) to gauge the need for additional fluid and ongoing resuscitation.
  Interventions: Device: CardioQ-EDM and CipherOx-CRI

INTERVENTIONS:
Device: CardioQ-EDM and CipherOx-CRI — A CardioQ-EDM probe will be placed on the day of surgery after induction of general anesthesia. The anesthesiologist will inform the investigator of plans to provide a fluid or blood bolus per clinical judgement in addition to the protocolized 10 ml/kg bolus provided after induction. While the anesthesiologist is preparing to administer volume expansion, a co-investigator will collect pre-fluid bolus data. Measurements will be recorded for data analysis at the completion of the trial. Additionally, a CipherOx-CRI probe will be placed on the patient's index finger (recorded data will be interpreted post hoc) and a bedside ultrasound will be performed by either the principal investigator (PI) or one of two co-investigators to measure the IVC CI. Ultrasound cine-loops will be recorded, and CI will be calculated post-hoc. Data will be recorded on the Data Collection Form for each fluid bolus administered. The PI and co-investigators will manage all aspects of investigational devices.

SUMMARY:
The goal if this study is to employ the CardioQ-Esophageal Aortic Doppler probe to define fluid responders from non-responders among infants undergoing cranial vault reconstruction for craniosynostosis. After defining these two groups in this single arm prospective trial, the investigators will compare the predictive utility of non-invasive devices such as the CipherOx-Compensatory Reserve Index (CipherOx-CRI) and Inferior Vena Cava Collapsibility Index (IVC CI) to currently employed indices (heart rate, systolic blood pressure, urine output and pulse pressure variability) to gauge the need for additional fluid and ongoing resuscitation. If the CipherOx-CRI or IVC CI proved to be as predictive or better at predicting fluid responders, the investigators hope to replace invasive arterial lines with non-invasive tools to guide resuscitation.

DETAILED DESCRIPTION:
Predicting fluid responsiveness in the operating room is essential to guide balanced resuscitation. Aggressive resuscitation may lead to significant morbidities, such as intra-abdominal hypertension, pulmonary edema, difficulty with ventilator liberalization, and consequently increased mortality. Alternatively, under resuscitation may lead to mal-perfusion and end-organ dysfunction.

A plethora of indices and tools have been studied and marketed to assess intravascular volume status with only a few proven reliable with reproducible results. Based on pre-fluid challenge values, several of these tools have been used to predict who may benefit from additional fluid (fluid responders). Alternatively, some of these tools have been used to distinguish fluid responders from non-responders based on changes in pre- and post-fluid challenge values. Among these tools, the pulmonary artery catheter provides measurements of both left and right heart pressures which can be applied to calculate the cardiac output (CO) and stroke volume (SV). Changes in these values (e.g. an increase in the stroke volume by 10%) between pre- and post-fluid challenge have been used to define fluid responders. This devise, however, is invasive with several significant risks, and therefore is rarely used in children. Echocardiography, on the other hand, is a non-invasive bedside study also used to assess CO and SV but is expensive and requires trained echosonagraphers for application. Further, because a transthoracic probe is required to obtain the images, application in the operating room is difficult as the chest is often in the operating field limiting access to the echosonagrapher. Lastly, the esophageal aortic blood flow device (CardioQ-Esophageal Dopler Monitor (Cardio-EDM), Deltex Medical, Chichester, UK) has been found in multiple adult and pediatric studies to reliably distinguish fluid responders from non-responders intensive care unit (ICU) and operating room. Much like an orogastric tube, this device is simply placed by a provider in the patient's esophagus and uses Doppler waveforms to measure aortic blood flow velocities. Variations in the amplitude of peak velocities has been shown to corelate with intravascular volume status. Specifically, a change in the peak velocity by greater than 10% between pre- and post-fluid challenge values has been shown to accurately distinguishes those who are fluid responsive from those who are not with similar accuracy to echocardiography and pulmonary artery catheter readings.

In recent years with continued technological advancements, there has been enthusiasm about less invasive, and in some cases, non-invasive, tools to gauge volume status. Among these, bedside ultrasonography (performed by providers rather than sonographers) is a common tool used to evaluate the inferior vena cava (IVC) collapsibility index (CI) has been shown to be a reliable tool in adults. Another non-invasive device uses a photoplethysmoraphic probe (CipherOx-CRI) placed on a digit to calculate the compensatory reserve index (CRI), a marker of proximity to hemodynamic collapse. Both IVC CI and CRI have been shown in multiple adult studies to predictive the need for volume expansion, but their utility in the pediatric population is unknown.

The goal if this proposed study is to employ the CardioQ-EDM probe to define fluid responders from non-responders among infants undergoing cranial vault reconstruction for craniosynostosis. After defining these two groups in this single arm prospective trial, the investigators will compare the predictive utility of non-invasive devices such as the CipherOx-CRI and IVC CI to currently employed indices (heart rate, systolic blood pressure, urine output and pulse pressure variability) to gauge the need for additional fluid and ongoing resuscitation. If the CipherOx-CRI or IVC CI proved to be as predictive or better at predicting fluid responders, the investigators hope to replace invasive arterial lines with non-invasive tools to guide resuscitation.

The investigators chose this population for several reasons. First, the investigators institution performs approximately 50-70 of these cases a year making them a relatively accessible group. Second, these children are generally healthy which will minimize physiologic confounders. Additionally, the subjects are paralyzed, have normal respiratory compliance, and providers maintain normothermia, all of which will minimizing confounders. Another unique benefit to this population is that these infants have been nil per os for several hours prior to surgery, putting them at risk for hypovolemia, and after induction, independent of the provider's assessment of intravascular volume status, all children receive a bolus of crystalloid (10mL/kg). This baseline data should provide sufficient data for analysis; but because these procedures are associated with significant blood loss and hypovolemia requiring aggressive resuscitation in the form of fluid or blood boluses, the investigators plan to continue to collect pre- and post- bolus data with the hope to further validate the benefit of non-invasive tools such as the CipherOx-CRI and IVC CI in the setting of ongoing blood loss.

As intravascular volume status is often difficult to assess clinically, the investigators aim to determine the predictability of non-invasive devices to guide resuscitation. In this prospective observational study, the investigators hope to identify:

1. The proportion of children within the cohort who are fluid responsive based on CardioQ-EDM aortic blood flow velocity changes pre- and post-bolus,
2. The positive predictive value, negative predictive value, sensitivity, specificity, and optimal threshold for CRI, IVC CI, pulse pressure variability, stroke volume variability, heart rate, systolic blood pressure, and mean arterial pressures in predicting fluid responders as determined by CardioQ-EDM, and
3. Assess confounding variables that may influence the predictive utility of such devices

ELIGIBILITY:
Inclusion Criteria:

* Children with craniosynostosis undergoing cranial vault reconstruction

Exclusion Criteria:

* Children with known underlying cardiac anomalies or cardiac arrhythmias
* Weight less than 3 kg
* Children who have vasopressors adjusted during a fluid bolus

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarkis Derderian, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers is planned

REFERENCES:
- [Background] Malbrain ML, Marik PE, Witters I, Cordemans C, Kirkpatrick AW, Roberts DJ, Van Regenmortel N. Fluid overload, de-resuscitation, and outcomes in critically ill or injured patients: a systematic review with suggestions for clinical practice. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):361-80. doi: 10.5603/AIT.2014.0060. PMID 25432556
- [Background] Feissel M, Michard F, Mangin I, Ruyer O, Faller JP, Teboul JL. Respiratory changes in aortic blood velocity as an indicator of fluid responsiveness in ventilated patients with septic shock. Chest. 2001 Mar;119(3):867-73. doi: 10.1378/chest.119.3.867. PMID 11243970
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Esophageal Doppler monitoring predicts fluid responsiveness in critically ill ventilated patients. Intensive Care Med. 2005 Sep;31(9):1195-201. doi: 10.1007/s00134-005-2731-0. Epub 2005 Jul 30. PMID 16059723
- [Background] Durand P, Chevret L, Essouri S, Haas V, Devictor D. Respiratory variations in aortic blood flow predict fluid responsiveness in ventilated children. Intensive Care Med. 2008 May;34(5):888-94. doi: 10.1007/s00134-008-1021-z. Epub 2008 Feb 8. PMID 18259726
- [Background] Absi MA, Lutterman J, Wetzel GT. Noninvasive cardiac output monitoring in the pediatric cardiac Intensive Care Unit. Curr Opin Cardiol. 2010 Mar;25(2):77-9. doi: 10.1097/HCO.0b013e3283362452. PMID 20104174
- [Background] Weber T, Wagner T, Neumann K, Deusch E. Low predictability of three different noninvasive methods to determine fluid responsiveness in critically ill children. Pediatr Crit Care Med. 2015 Mar;16(3):e89-94. doi: 10.1097/PCC.0000000000000364. PMID 25647238
- [Background] Pereira de Souza Neto E, Grousson S, Duflo F, Ducreux C, Joly H, Convert J, Mottolese C, Dailler F, Cannesson M. Predicting fluid responsiveness in mechanically ventilated children under general anaesthesia using dynamic parameters and transthoracic echocardiography. Br J Anaesth. 2011 Jun;106(6):856-64. doi: 10.1093/bja/aer090. Epub 2011 Apr 26. PMID 21525016
- [Background] Lanspa MJ, Grissom CK, Hirshberg EL, Jones JP, Brown SM. Applying dynamic parameters to predict hemodynamic response to volume expansion in spontaneously breathing patients with septic shock. Shock. 2013 Feb;39(2):155-60. doi: 10.1097/SHK.0b013e31827f1c6a. PMID 23324885
- [Background] Janak JC, Howard JT, Goei KA, Weber R, Muniz GW, Hinojosa-Laborde C, Convertino VA. Predictors of the Onset of Hemodynamic Decompensation During Progressive Central Hypovolemia: Comparison of the Peripheral Perfusion Index, Pulse Pressure Variability, and Compensatory Reserve Index. Shock. 2015 Dec;44(6):548-53. doi: 10.1097/SHK.0000000000000480. PMID 26529655
- [Background] Czerwinski M, Hopper RA, Gruss J, Fearon JA. Major morbidity and mortality rates in craniofacial surgery: an analysis of 8101 major procedures. Plast Reconstr Surg. 2010 Jul;126(1):181-186. doi: 10.1097/PRS.0b013e3181da87df. PMID 20220557
- [Background] Swan HJ, Ganz W, Forrester J, Marcus H, Diamond G, Chonette D. Catheterization of the heart in man with use of a flow-directed balloon-tipped catheter. N Engl J Med. 1970 Aug 27;283(9):447-51. doi: 10.1056/NEJM197008272830902. No abstract available. PMID 5434111
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wheeler AP, Bernard GR, Thompson BT, Schoenfeld D, Wiedemann HP, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Pulmonary-artery versus central venous catheter to guide treatment of acute lung injury. N Engl J Med. 2006 May 25;354(21):2213-24. doi: 10.1056/NEJMoa061895. Epub 2006 May 21. PMID 16714768
- [Background] Shah MR, Hasselblad V, Stevenson LW, Binanay C, O'Connor CM, Sopko G, Califf RM. Impact of the pulmonary artery catheter in critically ill patients: meta-analysis of randomized clinical trials. JAMA. 2005 Oct 5;294(13):1664-70. doi: 10.1001/jama.294.13.1664. PMID 16204666
- [Background] Sandham JD, Hull RD, Brant RF, Knox L, Pineo GF, Doig CJ, Laporta DP, Viner S, Passerini L, Devitt H, Kirby A, Jacka M; Canadian Critical Care Clinical Trials Group. A randomized, controlled trial of the use of pulmonary-artery catheters in high-risk surgical patients. N Engl J Med. 2003 Jan 2;348(1):5-14. doi: 10.1056/NEJMoa021108. PMID 12510037
- [Background] Westphal GA, Goncalves AR, Bedin A, Steglich RB, Silva E, Poli-de-Figueiredo LF. Vasodilation increases pulse pressure variation, mimicking hypovolemic status in rabbits. Clinics (Sao Paulo). 2010 Feb;65(2):189-94. doi: 10.1590/S1807-59322010000200011. PMID 20186303
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Chytra I, Pradl R, Bosman R, Pelnar P, Kasal E, Zidkova A. Esophageal Doppler-guided fluid management decreases blood lactate levels in multiple-trauma patients: a randomized controlled trial. Crit Care. 2007;11(1):R24. doi: 10.1186/cc5703. PMID 17313691
- [Background] Desgranges FP, Desebbe O, Pereira de Souza Neto E, Raphael D, Chassard D. Respiratory variation in aortic blood flow peak velocity to predict fluid responsiveness in mechanically ventilated children: a systematic review and meta-analysis. Paediatr Anaesth. 2016 Jan;26(1):37-47. doi: 10.1111/pan.12803. Epub 2015 Nov 6. PMID 26545173
- [Background] Zhao J, Wang G. Inferior Vena Cava Collapsibility Index is a Valuable and Non-Invasive Index for Elevated General Heart End-Diastolic Volume Index Estimation in Septic Shock Patients. Med Sci Monit. 2016 Oct 20;22:3843-3848. doi: 10.12659/msm.897406. PMID 27762259
- [Background] Preau S, Bortolotti P, Colling D, Dewavrin F, Colas V, Voisin B, Onimus T, Drumez E, Durocher A, Redheuil A, Saulnier F. Diagnostic Accuracy of the Inferior Vena Cava Collapsibility to Predict Fluid Responsiveness in Spontaneously Breathing Patients With Sepsis and Acute Circulatory Failure. Crit Care Med. 2017 Mar;45(3):e290-e297. doi: 10.1097/CCM.0000000000002090. PMID 27749318
- [Background] Gan H, Cannesson M, Chandler JR, Ansermino JM. Predicting fluid responsiveness in children: a systematic review. Anesth Analg. 2013 Dec;117(6):1380-92. doi: 10.1213/ANE.0b013e3182a9557e. PMID 24257389
- [Background] Muniz GW, Wampler DA, Manifold CA, Grudic GZ, Mulligan J, Moulton S, Gerhardt RT, Convertino VA. Promoting early diagnosis of hemodynamic instability during simulated hemorrhage with the use of a real-time decision-assist algorithm. J Trauma Acute Care Surg. 2013 Aug;75(2 Suppl 2):S184-9. doi: 10.1097/TA.0b013e31829b01db. PMID 23883906
- [Background] Stewart CL, Mulligan J, Grudic GZ, Convertino VA, Moulton SL. Detection of low-volume blood loss: compensatory reserve versus traditional vital signs. J Trauma Acute Care Surg. 2014 Dec;77(6):892-7; discussion 897-8. doi: 10.1097/TA.0000000000000423. PMID 25423536
- [Background] Monnet X, Bleibtreu A, Ferre A, Dres M, Gharbi R, Richard C, Teboul JL. Passive leg-raising and end-expiratory occlusion tests perform better than pulse pressure variation in patients with low respiratory system compliance. Crit Care Med. 2012 Jan;40(1):152-7. doi: 10.1097/CCM.0b013e31822f08d7. PMID 21926581
- [Background] Teboul JL, Monnet X, Chemla D, Michard F. Arterial Pulse Pressure Variation with Mechanical Ventilation. Am J Respir Crit Care Med. 2019 Jan 1;199(1):22-31. doi: 10.1164/rccm.201801-0088CI. PMID 30138573
- [Background] Airapetian N, Maizel J, Alyamani O, Mahjoub Y, Lorne E, Levrard M, Ammenouche N, Seydi A, Tinturier F, Lobjoie E, Dupont H, Slama M. Does inferior vena cava respiratory variability predict fluid responsiveness in spontaneously breathing patients? Crit Care. 2015 Nov 13;19:400. doi: 10.1186/s13054-015-1100-9. PMID 26563768
- [Background] Tibby SM, Hatherill M, Murdoch IA. Use of transesophageal Doppler ultrasonography in ventilated pediatric patients: derivation of cardiac output. Crit Care Med. 2000 Jun;28(6):2045-50. doi: 10.1097/00003246-200006000-00061. PMID 10890662

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluid Challenge Responders: This arm was defined as those who had an increase in their peak aortic velocity of > 15% measured by the CardioQ-Esophageal Doppler Monitor following a crystalloid bolus (10 mL/kg)
- Fluid Challenge Non-responders: This arm was defined as those who did not have an increase in their peak aortic velocity of > 15% measured by the CardioQ-Esophageal Doppler Monitor following a crystalloid bolus (10 mL/kg)
Period: Overall Study
Arm/Group | Fluid Challenge Responders | Fluid Challenge Non-responders
Started | 7 | 16
Completed | 7 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Challenge Responders | Fluid Challenge Non-responders | Total
Number analyzed (Participants) | 7 | 16 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 16 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 12 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 14 | 19
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 13 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 16 | 23

OUTCOME MEASURES:

1. Primary Outcome: Utility of Compensatory Reserve Index (CRI) Which Ranges From 0-1 in Order to Predict Fluid Responders From Non-responders
Description: Using a delta peak aortic velocity threshold of 10% (measured from CardioQ-EDM) before and after a bolus to define fluid responders (=/>10%) from non-responders (<10%), we will determine the performance of pre-bolus CRI reading which is an index between 0 and 1 (0=poor reserve and 1=excellent reserve) in order to predict fluid responders from non-responders. Measurements will be recorded three times with one minute between measurements and then averaged.
  Vital signs analyzed included heart rate, systolic blood pressure, mean arterial pressure, shock index (heart rate/systolic blood pressure), pulse pressure variability, and end-tidal carbon dioxide level. Infants were also monitored with a Compensatory Reserve Index (CRI) monitor, which provides a continuous, individual-specific, beat-to-beat estimate of central volume status, from normovolemia (CRI=1) to decompensation (CRI=0). Each variable's performance was compared using area under the receiver operator curves (AUC).
Time Frame: Through study completion (3-4 hours)
Population: Fluid responders vs non-fluid responders
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluid Challenge Responders | Fluid Challenge Non-responders
Number analyzed (Participants) | 7 | 16
units on a scale | 0.06 (0.03) | 0.05 (0.02)

ADVERSE EVENTS:
Time Frame: Data was collected from the time of probe placement in the operating room until discharge (0-3 days)
Arm/Group | Fluid Challenge Responders | Fluid Challenge Non-responders
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/16
Other Adverse Events (participants affected / at risk) | 0/7 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03915587/Prot_SAP_000.pdf